CLINICAL TRIAL: NCT02113176
Title: Minocycline as Neuroprotectant After Aneurysmal Subarachnoid Hemorrhage
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding of minocycline
Sponsor: University at Buffalo (Other)
Collaborators: University at Buffalo Neurosurgery (Other)
Responsible Party: Principal Investigator, Adnan H. Siddiqui, Associate Professor of Neurosurgery & Radiology, Director of Neurosurgical Research, Director of Stroke Service, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MINO-SAH
Record Dates: First submitted 2014-01-31; First posted 2014-04-14 (Estimated); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Subarachnoid Aneurysm Hemorrhage
Keywords: SAH
MeSH Terms: interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline (Experimental): * 200 mg IV/placebo
  * Followed by 100 mg IV BID x 7days
  * Followed by 200 mg tablet QD x 14days
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): 200 mg IV/placebo
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline

SUMMARY:
The purpose of this study is to determine the safety and efficacy of a drug minocycline in improving outcomes at 3 months after rupture of an aneurysm in the head.

DETAILED DESCRIPTION:
Prior to the drug:

If you decide to take part in this study, you will have a brief interview about your medical history and any medications you are taking. You will have a medical and neurological examination, CT scan and/or an angiogram to look at the blood vessel and blood supply going to the brain, and blood samples drawn for a complete blood count, chemistry analysis and cardiac enzymes (to assess any recent damage to your heart). You will have a surgery or an image guided procedure to close your aneurysm.

Additionally, during the course of the study you may be asked to have a computerized tomography (CT scan) or magnetic resonance imaging (MRI) if there is a necessity. These tests will reveal areas that might have been damaged in your brain.

Drug:

If the tests show that you qualify as a candidate for this study, you will be randomly assigned (like a flip of a coin) to have either the minocycline drug or a dummy drug that looks the same but does not have the drug in it. For the first 7 days, the drug will be given as an injection two times a day and after that for 14 days once a day by mouth. Rest of the care will be standard like in any aneurysm patient. We study the status of your blood vessel surrounding the brain with ultrasound daily to see if they have any narrowing. If the doctors find any narrowing, you will be treated to relive the narrowing. If you are discharged home at any point in the 21 days, you will be switch the oral drug and given the required drugs with instructions.

Follow up:

Before you are discharged from the hospital and at 7, 21, 30 and 90 days after the start of the drug, the following evaluations will be performed: a complete physical and neurological examinations.

As part of this study, you are required to return to the hospital or to your physician at one (1), seven (7), twenty-one (21), thirty (30), ninety (90) days after stroke onset. You will have a physical exam, a complete neurological exam. Additionally, you will be asked questions about any health problems or hospitalizations you have had since you were discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 yrs of age
* Ruptured aneurysm
* Initiate treatment within 72 hours of SAH
* Pre Rankin ≤ 1

Exclusion Criteria:

* Hunt & Hess 5 with no improvement
* ICP > 30
* No plans to treat aneurysm
* Allergy to Tetracycline / Antibiotics
* Creatinine >2
* Platelets < 75,000
* Other brain diseases
* Previous infection requiring Tetracycline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
adverse event | 21 days
  The primary objective of the study is to evaluate the effectiveness of minocycline in improving outcomes for patients after aneurysmal SAH.
  To determine the safety of minocycline 200mg/day for 21 days in the treatment arm after aneurysmal subarachnoid hemorrhage.

SECONDARY OUTCOMES:
comparative stroke scale | 3 months
  To demonstrate a significant difference in outcome at 3 months as measured by NIHSS, mRS, BI and GOS in the minocycline treatment group when compared to the placebo arm.
  To determine any significant differences in vasospasm rates, duration of vasospasm, interventions for vasospasm, vasospasm related infarcts and delayed ischemic deficits between minocycline and placebo arms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Buffalo Neurosurgery, Buffalo, New York, United States